CLINICAL TRIAL: NCT01702883
Title: Using an Internet Survey to Improve Patient Adherence in Chronic Disease
Brief Title: The Medication Experience Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: IRB00020789
Record Dates: First submitted 2012-10-04; First posted 2012-10-10 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2025-04

CONDITIONS: Hypertension; Elevated Cholesterol; Diabetes; Depression
Keywords: prescriptions; hypertension; high cholesterol; diabetes; depression; adherence
MeSH Terms: conditions — Hypertension; Hypercholesterolemia; Diabetes Mellitus; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Randomization occurs after enrollment survey has been completed. This group will not receive the internet intervention for the twelve months. They will be asked to complete the final survey.
- Intervention Group A (Experimental): Randomization occurs after enrollment survey has been completed. Upon secondary randomization at week eight, this group will continue to receive weekly internet surveys for the entire twelve months. They will be asked to complete the final survey.
  Interventions: Other: Internet Survey
- Intervention Group B (Experimental): Randomization occurs after enrollment survey has been completed. This group will complete weekly internet surveys for eight weeks. Upon secondary randomization at week eight, this group will begin to receive monthly internet surveys. They will be asked to complete the final survey.
  Interventions: Other: Internet Survey
- Intervention Group C (Experimental): Randomization occurs after enrollment survey has been completed. This group will complete weekly internet surveys for eight weeks. Upon secondary randomization at week eight, the group will not receive any more internet surveys. They will be asked to complete the final survey.
  Interventions: Other: Internet Survey

INTERVENTIONS:
Other: Internet Survey — prompt to complete internet survey
  Other Names: internet surveys
  Arms: Intervention Group A; Intervention Group B; Intervention Group C

SUMMARY:
The purpose of this study is to evaluate whether participation in an Internet-based intervention helps improve medication use.

ELIGIBILITY:
Inclusion Criteria:

* Any male or female 18 years or older, filling prescriptions for oral medications for hypertension, high cholesterol, diabetes, or depression at the Downtown Health Plaza, Piedmont Plaza, or Cancer Center Pharmacies.

Exclusion Criteria:

* Inability to complete Internet surveys due to inadequate Internet access, not understanding a survey written in English, or lack of computer skills.
* Patient does not intend to continue using the same WFBMC-affiliated pharmacy for the next 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2012-10; Primary Completion 2015-07-31 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
The primary measure will be adherence as measured by pharmacy refills in each group. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Steve R Feldman, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

DOCUMENTS (1):
  • Informed Consent Form (2014-07-16): https://cdn.clinicaltrials.gov/large-docs/83/NCT01702883/ICF_000.pdf